CLINICAL TRIAL: NCT03254771
Title: Effectiveness of a Decision Aid for Patients With Knee Osteoarthritis Candidates for Primary Total Arthroplasty
Brief Title: Effectiveness of a Decision Aid for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: Hospital de Basurto (Other); Hospital Donostia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PI15-01264
Record Dates: First submitted 2017-06-05; First posted 2017-08-18 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Knee ostheoartritis; Arthroplasty; Clinical trial; Decision aids
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Decision Support Techniques

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): In the control group, the usual explanation about the disease and the possibilities of treatment will be followed
- Intervention group (Experimental): In the Intervention group, the Decision Aid (DA) will be presented and explained to the patient by research personnel at a schedule previously agreed with the patient. The patient will be given a paper copy of the (DA) to take home, as well as a web link to the computer application, and oral and written instructions to review the material again and perform value clarification exercises.
  Interventions: Other: Decision aid

INTERVENTIONS:
Other: Decision aid — Decision aids are tools that enables to promote and facilitate patients' involvement in medical decisions concerning their health
  Arms: Intervention group

SUMMARY:
The main goal of this study is assess the effectiveness of a DA for patients with knee osteoarthritis candidates to ART

DETAILED DESCRIPTION:
The number of knee total arthroplasty (ART) interventions has increased in the last 10 years in European countries, partly due to the aging of the population and partly because of the increase in the use of these interventions to improve the quality of life among elderly patients. According to the Organization for Economic Cooperation and Development (OECD) 2012, from 2000 to 2010 in Spain the percentage of knee ART has doubled in recent years. .

The role of citizens in decisions affecting their health is changing. Individual factors such as improving educational attainment and access to medical information, and collective factors such as training of patient groups and changes in legislation (informed consent, autonomy principle) have motivated the transition from a paternalistic model to a co-responsibility model. Shared decision-making (TDC) has been proposed in recent years as a model of care that promotes users' involvement in the decisions about their treatment, in those situations where there is uncertainty and / or the scientific evidence reports a balance between benefits and risks that is similar for two or more therapeutic options. Decision aids (DA) are tools designed to promote and facilitate patients' involvement in medical decisions concerning their health

Objectives:

To assess the effectiveness of a DA for patients with knee osteoarthritis candidates to ART

Methodology:

Randomized controlled trial to evaluate the effectiveness of the DA versus usual care in reducing decisional conflict, increasing knowledge of the disease/treatments, informed choice and the satisfaction with the decision making process, and decreasing decisional regret.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis of the knee
* Candidates for arthroplasty

Exclusion Criteria:

* Patients who have already undergone knee arthroplasty
* Patients younger than 18 years

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2017-08-16 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Decisional conflict, measured by the Decisional Conflict Scale (DCS). | Immediately after the intervention; 6 months after the intervention (only non-operated patients)
  The DCS measures patients' uncertainty about treatment choice. It is composed of five subscales: uninformed, values, support, uncertainty and effectiveness

SECONDARY OUTCOMES:
Knowledge of the disease and treatments | Immediately after the intervention; 6 months after the intervention (only non-operated patients)
  A 7-item scale will be udes to assess patients' knowledge of the disease and treatments
Goals and concerns | Immediately after the intervention; 6 months after the intervention (only non-operated patients)
  A 10-item scale will assess the importance that patients attribute to different characteristics of avaliable treatments
Treatment preference | Immediately after the intervention; 6 months (only non-operated patients)
  Patients will be asked the treatment they prefer: AINEs, knee injections or arthroplasty
Satisfaction with the decision making process | Immediately after the intervention; 6 months
  The scale developed by Barry et al. (1997) will be used, composed of 12 items measuring patients' satisfaction with information and care provided
Decisional regret, measured by the Decisional Regret Scale (DRS) | 6 months (only operated patients)
  The DRS contains five items measuring patients regret with the treatment decision

CONTACTS AND LOCATIONS:
Overall Officials: Amado Rivero Santana, PhD, Study Chair — Researcher
Locations (1):
- Servicio de Evaluación de. Servicio Canario de Salud -, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No